CLINICAL TRIAL: NCT06682832
Title: Comparison of Exercise Capacity, Muscle Strength and Oxygenation, Arterial Stiffness, Physical Activity and Quality of Life in Individuals with Chronic Obstructive Pulmonary Disease and Impaired Spirometry with Preserved Ratio
Brief Title: Comparison of Clinical Status of Individuals with COPD and Preserved Ratio Impaired Spirometry
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ece Kumlu, Principal Investigator, Hacettepe University
Other Study IDs: HU-FTR-KUMLUE-01
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Preserved Ratio Impaired Spirometry (PRISM)
Keywords: COPD; PRISm; exercise capacity; muscle strength; arterial stiffness; physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- COPD group: Consisted of 18 individuals over 40 years of age with chronic obstructive pulmonary disease.
- PRISm group: Consisted of 18 individuals over 40 years of age with preserved ratio impaired spirometry.
- Healthy group: Consisted of 18 healthy individuals over 40 years of age.

SUMMARY:
Despite the globally varying high prevalence rate of the PRISm phenotype, there are no guidelines for its diagnostic evaluation and management. Further studies are needed on appropriate approaches for individuals with PRISm to improve respiratory symptoms and prognosis. As research continues to evolve, PRISm needs to be recognized as a critical component of pulmonary assessments and at-risk individuals need to be provided with appropriate treatment and follow-up to prevent progression to COPD. There are no studies in the literature comparing PRISm, respiratory muscle strength, peripheral muscle strength and oxygenation, arterial stiffness, physical activity level and sleep level in COPD and healthy individuals. The aim of this study was to compare respiratory muscle strength, peripheral muscle strength and oxygenation, arterial stiffness, physical activity level and sleep level in PRISm, COPD and healthy subjects.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common, preventable and treatable multisystemic lung disease characterised by chronic respiratory symptoms (dyspnoea, cough, expectoration and/or exacerbations) due to abnormalities in the airways causing permanent and often progressive airflow limitation. In a part of the individuals with affected lung function, FEV1/FVC is preserved after bronchodilation (≥ 70%), whereas FEV1 is lower than expected (< 80%). This condition, which describes a preserved ratio impaired spirometry (PRISm), is highly prevalent in current and former smokers. PRISm is defined as a spirometry pattern that is not always a stable phenotype, but should be considered ''patient'' because symptoms and/or functional and/or structural abnormalities are present and therefore require care and treatment. There are studies showing that pulmonary functions, exercise capacity and quality of life are impaired in individuals with PRISm, whose pathophysiology is unclear and clinical effects are not known. In addition to the insufficient number of studies investigating exercise capacity, quality of life and pulmonary function on behalf of PRISm in the literature, no previous studies comparing respiratory muscle strength, peripheral muscle strength and oxygenation, arterial stiffness, physical activity level and sleep level in PRISm, COPD and healthy individuals have been found. In this study, aimed to investigate whether the parameters (symptoms, respiratory and peripheral muscle strength, physical activity level, exercise capacity, muscle oxygenation, arterial stiffness), which have been proven to be affected in the COPD group due to their clinical similarity with COPD, are affected in the PRISm group. A total of 54 individuals, 18 in each group, will be included in the study. Pulmonary function, symptoms, body composition, respiratory muscle strength, peripheral muscle strength, exercise capacity, tissue oxygenation, arterial stiffness, physical activity levels, sleep and quality of life will be compared in PRISm, COPD and healthy individuals. Our study will be able to reveal the clinical status of PRISM patients in terms of pulmonary function, symptoms, body composition, respiratory muscle strength, peripheral muscle strength, exercise capacity, tissue oxygenation, arterial stiffness, physical activity levels, sleep and quality of life compared to COPD group and healthy group and will be a guide in planning pulmonary rehabilitation programmes.

ELIGIBILITY:
Inclusion Criteria:

PRISm group inclusion criteria;

* Being >40 years old,
* Being diagnosed with PRISm,
* Volunteering to participate in the study,
* Not having any orthopaedic or neurological problems that may prevent participation in the measurements,
* Co-operation with measurements

Inclusion criteria for the COPD group;

* Being >40 years old,
* Being diagnosed with COPD,
* To be clinically stable,
* Volunteering to participate in the study.

Inclusion criteria for healthy individuals;

* Being >40 years old,
* Volunteering to participate in the study,
* No known chronic health problems,
* To be able to co-operate with the measurements.

Exclusion Criteria:

PRISm group exclusion criteria;

* Being diagnosed with COPD,
* Severe orthopaedic, neurological and cardiac diseases
* Not volunteering to participate in the study

Exclusion criteria for COPD group;

* Severe orthopaedic, neurological and cardiac diseases,
* Being in COPD exacerbation period,
* Not volunteering to participate in the study.

Healthy individuals exclusion criteria;

* Having a known chronic disease,
* Not volunteering to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD and PRISm patients referred to the Cardiopulmonary Rehabilitation Unit for routine physiotherapy and rehabilitation will be included in the study. The group of healthy individuals will be formed by including the healthy siblings of the participants who are age and gender compatible with the COPD and PRISm groups, and the volunteers among the relatives and acquaintances of the researchers. 54 individuals will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 6 minutes
  Exercise capacity is assessed using the 6-minute walk test (6MWT). The 6MWT is performed according to the criteria of the American Thoracic Society.
Arterial Stiffness | 20 minutes
  Arterial stiffness is evaluated with a Tel-O-Graph CT device with oscillometric cuff (I.E.M., Stolberg, Germany). Central systolic blood pressure, pulse wave velocity (PWV) and augmentation index (Alx) are measured with brachial pulse waves. After a five-minute rest, three measurements are performed in a quiet environment.
Muscle Oxygenation | 10 minutes
  Muscle oxygenation is assessed using a measurement and monitoring device (Moxy Fortiori Design LLC, Minnesota, USA). The device is placed on the vastus lateralis muscle. Resting measurements are taken for at least 3 minutes until the muscle oxygen saturation (SmO2) signal stabilizes. SmO2 at rest, SmO2 during 6DYT and during the first minute of recovery, and mean SmO2 are recorded.
Physical Activity | 5 minutes
  Physical activity levels is assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). The IPAQ requires respondents to estimate time spent in various levels of physical activity during the previous week. Scores for walking and moderate and vigorous activities are calculated as durations and frequencies multiplied by known metabolic equivalents per activity. The results for all activity-based items are summed for the total physical activity score. The participants were then categorized as inactive, minimally active and sufficiently active according to the IPAQ categorical classification.

SECONDARY OUTCOMES:
Body Composition | 5 minutes
  Body composition is evaluated by Bioelectrical Impedance Analysis method. For body composition measurement, it is completed in an upright posture, without moving, leaving a space between the arms and torso, ensuring full contact of the hands and feet with the electrodes. Muscle mass, fat mass, body fat percentage (BMR) and lean body weight (LBW) values of the participants are recorded.
Respiratory Muscle Strength | 10 minutes
  Respiratory Muscle Strength is measured using a mouth pressure meter (MicroRPM, Micro Medical, Rochester, UK) and personalized antibacterial and antiviral disposable filters; maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) values are determined.
Peripheral Muscle Strength | 5 minutes
  Peripheral muscle strength is measured by knee extensor muscle strength measurement. Measurements are performed with a portable digital muscle strength measuring device (01165 Manual Muscle Tester, Lafayette Instrument Co. Lafayette, USA).
Sleep Quality | 5 minutes
  Sleep quality is measured by the Pittsburgh Sleep Quality Index (PSQI). The scale assesses sleep quality and sleep disturbance over the past month. The scale includes 24 questions. The total PDQI score ranges from 0-21 points. A total score greater than 5 points indicates "poor sleep quality".
COPD Assessment Test | 5 minutes
  The COPD Assessment Test, COPD Assessment Test Questionnaire (CAT), is an eight-item self-reported scale scored on a 0-5 point scale to assess symptoms associated with COPD. As a clinical impact, a total score of less than 10 points is interpreted as few symptoms, while a score of more than 10 points is interpreted as more symptoms.
Quality of Life | 10 minutes
  Quality of Life will be assessed with the St George Respiratory Questionnaire (SGRQ). SGRQ is a 76-item health-related quality of life assessment questionnaire.
Symptoms | 8 minutes
  Symptoms, dyspnea and fatigue level are assessed. Dyspnea is assessed with the modified Medical Research Council (mMRC) dyspnea scale. Fatigue levels of individuals will be assessed using the Fatigue Severity Scale (FSS).
Pulmonary Function Test (forced vital capacity (FVC)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses forced vital capacity (FVC). FVC is the volume of air exhaled with rapid and forceful exhalation following deep inspiration.
Pulmonary Function Test (forced expiratory volume in the first second (FEV1)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses forced expiratory volume in the first second (FEV1). Forced vital capacity is the volume of air removed in the first second from the start of the maneuver.
Pulmonary Function Test (FEV1/FVC) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses FEV1/FVC.
Pulmonary Function Test (peak flow rate (PEF)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses peak flow rate (PEF). PEF is measured by maximal inspiration followed by maximal exhalation maneuver.
Pulmonary Function Test (forced expiratory flow from 25-75% (FEF25-75%)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses forced expiratory flow from 25-75% (FEF25-75%). FEF25-75% mean flow rate at 50% of the forced vital capacity maneuver.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No